CLINICAL TRIAL: NCT04785430
Title: Incarceration Risk Factors in Inguinal Hernia.Prospective Observational Clinical Trial.
Brief Title: Incarceration Risk Factors in Inguinal Hernia.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Turgut Donmez, Bakirkoy EAH, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: BakirkoyEAH Hande1
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Incarcerated Inguinal Hernia; Strangulated Inguinal Hernia; Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who underwent elective inguinal hernia surgery: Patients who have applied to the general surgery outpatient clinic of Bakırköy Dr Sadi Konuk Training and Research Hospital, diagnosed with inguinal hernia and underwent hernia repair surgery.
- Patients who underwent emergency inguinal hernia surgery: Patients who have applied to the emergency clinic of Bakırköy Dr Sadi Konuk Training and Research Hospital, diagnosed with incarcerated inguinal hernia and underwent hernia repair surgery.

SUMMARY:
It is known that strangulation or necrosis of the intestine within the hernia sac of inguinal hernia increases mortality and morbidity in patients. However, the risks of incarceration in hernias have not been fully revealed.To better understand the factors associated with incarceration in inguinal hernia, the investigators will examine patients who will apply to our clinic for inguinal hernia and undergo elective and emergency inguinal hernia surgery.

DETAILED DESCRIPTION:
A prospective study will be conducted for 2 years, involving all adult patients who have applied to the general surgery outpatient clinic of Bakırköy Dr Sadi Konuk Training and Research Hospital, diagnosed with inguinal hernia, and who have applied to the emergency diagnosed with incarcerated inguinal hernia and underwent hernia repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-80
* Primary and recurrent inguinal hernias
* Incarcerated / strangulated inguinal hernias

Exclusion Criteria:

* Younger than 18, older than 80
* Pregnancy
* Mental retardation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have applied to the general surgery outpatient clinic of Bakırköy Dr Sadi Konuk Training and Research Hospital, diagnosed with inguinal hernia, and who have applied to the emergency diagnosed with incarcerated inguinal hernia and underwent hernia repair surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Hernia defect size | 2 hours after physical examination
  Measurement of fascial defect causing the hernia, using USG or CT

SECONDARY OUTCOMES:
Constipation | 1 years
  Frequent episodes without defecation lasting more than 3 days
Age | up to 24 weeks
  Patients age
Body Mass Index | up to 24 weeks
  Patients weight in kilograms divided by the square of height in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Donmez, Study Director — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakırkoy Dr.Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Sneiders D, Yurtkap Y, Kroese LF, Kleinrensink GJ, Lange JF, Gillion JF; Hernia-Club Members. Risk Factors for Incarceration in Patients with Primary Abdominal Wall and Incisional Hernias: A Prospective Study in 4472 Patients. World J Surg. 2019 Aug;43(8):1906-1913. doi: 10.1007/s00268-019-04989-x. PMID 30980102
- [Background] Kunduz E, Sormaz IC, Yapalak Y, Bektasoglu HK, Gok AF. Comparison of surgical techniques and results for emergency or elective femoral hernia repair. Ulus Travma Acil Cerrahi Derg. 2019 Nov;25(6):611-615. doi: 10.14744/tjtes.2019.04524. PMID 31701494
- [Derived] Kandemir H, Donmez T, Surek A, Gumusoglu AY, Karabulut M, Canoz O, Kaya A. Risk factors for incarceration in groin hernia: a prospective observational study. Hernia. 2025 Apr 12;29(1):142. doi: 10.1007/s10029-025-03331-w. PMID 40216639